CLINICAL TRIAL: NCT01106898
Title: A Phase II Study of Adjuvant Therapy Using a Regimen of Cyclophosphamide, Paclitaxel With or Without Trastuzumab in Stage I-II Breast Cancer Patients
Brief Title: Cyclophosphamide and Paclitaxel With or Without Trastuzumab in Stage I-II Breast Cancer Who Have Undergone Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0371-09-FB; NCI-2010-00608 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 371-09 (Other: University of Nebraska Medical Center); P30CA036727 (NIH)
Record Dates: First submitted 2010-04-13; First posted 2010-04-20 (Estimated); Results first posted 2018-05-31 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Stage IA Breast Cancer; Stage IB Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Paclitaxel; Taxes; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (chemotherapy with or without maintenance therapy) (Experimental): SYSTEMIC CHEMOTHERAPY: Patients receive cyclophosphamide IV over 1 hour and paclitaxel IV over 3 hours on day 1. Treatment repeats every 14 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY (Her-2 neu positive patients): Patients receive trastuzumab IV over 30 minutes on day 1. Treatment repeats every 14 days for 5 courses and then every 21 days for 14 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cyclophosphamide; Drug: paclitaxel; Biological: trastuzumab; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Biological: trastuzumab — Given IV
  Other Names: anti-c-erB-2; Herceptin; MOAB HER2
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies the side effects and how well giving cyclophosphamide and paclitaxel with or without trastuzumab works in treating patients with stage I-II breast cancer who have undergone surgery. Drugs used in chemotherapy, such as cyclophosphamide and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving monoclonal antibody therapy, such as trastuzumab, with chemotherapy may kill more tumor cells. Giving these treatments after surgery may kill any tumor cells that remain after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the toxicities and ability to complete the planned treatment of a dose-dense regimen of cyclophosphamide and paclitaxel with or without trastuzumab in patients with newly diagnosed stage I-II breast cancer.

II. To estimate recurrence free survival of a dose-dense regimen of cyclophosphamide and paclitaxel with or without trastuzumab in patients with newly diagnosed stage I-II breast cancer.

OUTLINE:

SYSTEMIC CHEMOTHERAPY: Patients receive cyclophosphamide intravenously (IV) over 1 hour and paclitaxel IV over 3 hours on day 1. Treatment repeats every 14 days for 6 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY (human epidermal growth factor receptor 2 [Her-2] neu positive patients): Patients receive trastuzumab IV over 30 minutes on day 1. Treatment repeats every 14 days for 5 courses and then every 21 days for 14 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed newly diagnosed stage I-II breast cancer
* Women of reproductive potential must be non-pregnant and non-nursing and must agree to employ an effective barrier method of birth control throughout the study and for up to 6 months following treatment
* Women of child-bearing potential must have a negative pregnancy test within 7 days of initiating study
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Absolute neutrophil count greater than or equal to 1,500/mcl
* Platelet count equal to or greater than 150,000/mcl
* Hemoglobin > 11 gm/dl
* Alkaline phosphatase equal or less than 1.5 times the upper limit of normal (ULN)
* Total bilirubin equal to or less than 1.5 times the ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) no greater than 1.5 times the ULN
* Creatinine less than 1.5 times the ULN
* Able to give informed consent
* All included patients must have normal cardiac function as defined by an ejection fraction of > 50% by echocardiogram
* Able to return for treatment and follow-up on the specified days

Exclusion Criteria:

* Prior malignancy; except for adequately treated basal cell or squamous cell skin cancer or noninvasive carcinomas
* Patients with preexisting grade II peripheral neuropathy
* Patients with prior chemotherapy
* Stage IV or metastatic breast cancer
* Pregnant or nursing women
* Inability to cooperate with treatment protocol
* No active serious infections or other conditions precluding chemotherapy
* Any comorbidity or condition which, in the opinion of the investigator, may interfere with the assessments and procedures of this protocol (e.g. unstable angina, myocardial infarction within 6 months, severe infection, etc.)
* Known hypersensitivity to any component of required drugs in the study
* Known positive for human immunodeficiency virus (HIV) or infectious hepatitis, type A, B or C or active hepatitis
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) class III or IV heart failure uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities; prior to study entry, any electrocardiograph (ECG) abnormality at screening has to be documented by the investigator as not medically relevant

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2010-03-24 (Actual); Primary Completion 2015-09-28 (Actual); Study Completion 2015-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth C Reed, Principal Investigator — University of Nebraska
Locations (2):
- United States (2):
  - Saint Francis Medical Center, Grand Island, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 112 subjects consented for this study, 3 were ineligible, 9 withdrew before study treatment starting. Only 100 subjects treated were available for analysis.
Groups:
- Treatment (Chemotherapy With or Without Maintenance Therapy): SYSTEMIC CHEMOTHERAPY: Patients receive cyclophosphamide IV over 1 hour and paclitaxel IV over 3 hours on day 1. Treatment repeats every 14 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY (Her-2 neu positive patients): Patients receive trastuzumab IV over 30 minutes on day 1. Treatment repeats every 14 days for 5 courses and then every 21 days for 14 courses in the absence of disease progression or unacceptable toxicity.
  cyclophosphamide, paclitaxel, trastuzumab: Given IV
Period: Overall Study
Arm/Group | Treatment (Chemotherapy With or Without Maintenance Therapy)
Started | 100
Completed | 94
Not Completed | 6
Not completed — Adverse Event | 6

BASELINE CHARACTERISTICS:
Population: Of the 112 subjects consented for this study, 3 were ineligible, 9 withdrew before study treatment starting. Only 100 subjects treated were available for analysis.
Arm/Group | Treatment (Chemotherapy With or Without Maintenance Therapy)
Number analyzed (Participants) | 112
Age, Continuous [Mean (Full Range); unit: years] | 57 [34 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 107
  Black, not of hispanic origin | 4
  Hispanic | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 112

OUTCOME MEASURES:

1. Primary Outcome: Recurrence-free Survival
Description: Recurrence-free survival curves will be plotted for subjects treated with stage I and II disease.
Time Frame: Time from the start of treatment to recurrence, second malignancy, or death as a first event, assessed up to 3 years
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Treatment (Chemotherapy With or Without Maintenance Therapy)
Number analyzed (Participants) | 100
percentage of subjects | 98 [92.2 to 99.5]

ADVERSE EVENTS:
Time Frame: Adverse events are collected from time the subject signs consent and ending 4 weeks following final chemotherapy (16 weeks for those not taking trastuzumab, Her-2 neu positive (add trastuzumab) patients this is 56 weeks). All subjects were also followed for only neuro and cardio toxicities for up to 3 months after final chemotherapy.
Description: Grade 3 and higher are reported per the CTC version 3.0 Number of participants for adverse event reporting is out of 102 patients because per the protocol every patient who fulfills all aspects of patient eligibility who receives a partial or complete course of chemotherapy will be evaluable for toxicity. There were 2 patients who started treatment and were removed from the study after 1 cycle due to adverse events.
Arm/Group | Treatment (Chemotherapy With or Without Maintenance Therapy)
All-Cause Mortality (participants affected / at risk) | 6/102
Serious Adverse Events (participants affected / at risk) | 16/102
Other Adverse Events (participants affected / at risk) | 57/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy With or Without Maintenance Therapy) (N=102)
Anaphylaxis (Immune system disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
thromboembolic event (Vascular disorders) | 2 (2) — pulmonary emboli and embolism
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 (3)
Skin Infection (Infections and infestations) | 1 (1) — cellulitis
Wound complication (Injury, poisoning and procedural complications) | 1 (1) — implant removed
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Duodenal perforation (Gastrointestinal disorders) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Infections and Infestations - Other (Infections and infestations) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2)
Lung infection (Infections and infestations) | 1 (1) — pneumonia
SinusTachycardia (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy With or Without Maintenance Therapy) (N=102)
Lymphocyte count decreased (Investigations) | 8 (12)
Hyperglycemia (Metabolism and nutrition disorders) | 23 (31)
Neutrophil count decreased (Investigations) | 14 (29)
Bone pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Nervous system disorders - Other (Nervous system disorders) | 7 (7) — neuropathy, unspecified
White blood cells decreased (Investigations) | 9 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes